CLINICAL TRIAL: NCT01551199
Title: Exposure Therapy for Veterans With PTSD and Panic Attacks (Phase 1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDA2-012-09F-1
Record Dates: First submitted 2012-03-02; First posted 2012-03-12 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: PTSD; Panic Attacks
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Panic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multiple Channel Exposure Therapy (Experimental): MCET-V is a cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks
  Interventions: Behavioral: Multiple Channel Exposure Therapy- Veterans

INTERVENTIONS:
Behavioral: Multiple Channel Exposure Therapy- Veterans — Individual therapy design completed over a 12-week period. The treatment will include psychoeducation about panic attacks and trauma and behavioral and cognitive exposure exercises.
  Other Names: MCET-V

SUMMARY:
To evaluate the feasibility, acceptability and effectiveness of Multiple Channel Exposure Therapy-Veterans (MCET-V) as a treatment for returning service members with comorbid posttraumatic stress disorder (PTSD) and panic disorder (PD) in two phases. The first phase of the study will examine the feasibility and acceptability of MCET-V.

DETAILED DESCRIPTION:
With the increasing number of Operations Iraqi Freedom and Enduring Freedom (OIF/OEF) veterans returning from war-zone areas, many will experience anxiety disorders such as PTSD and comorbid problems. Currently, about one in every six OIF/OEF veterans experiences PTSD and co-occurring PD. Although effective treatments exist for treating one or the other, we do not yet have treatments that can simultaneously target PTSD and PD. Thus, recent attention has focused on the development of multi-component treatments that simultaneously address PTSD and PD. This study is the first systematic investigation of a time-limited, multi-component cognitive-behavioral treatment for veterans with specific comorbid anxiety problems. The purpose of the first phase of the study is to evaluate the feasibility and acceptability of the multi-component cognitive-behavioral treatment in an open trial.

ELIGIBILITY:
Inclusion Criteria:

* being a veteran of any era;
* being enrolled in the Trauma Recovery Program (TRP) at the Michael E. DeBakey Veterans Affairs Medical Center (MEDVAMC), with a current diagnosis of PTSD and PD;
* being stable on psychotropic medication for 4 weeks before study participation; and
* being at least 18 years of age.

Exclusion Criteria:

* active substance dependence, or bipolar or psychotic disorders;
* severe depression and active suicidal ideation and intent (based on Structured Clinical Interview for DSM-IV disorders [SCID-IV] & Beck Depression Inventory-2nd edition [BDI-II]);
* cognitive impairment as indicated by the St. Louis University Mental Status exam (SLUMS); and
* veterans currently receiving psychosocial treatment specifically targeting PTSD or panic symptoms.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Teng, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Channel Exosure Therapy (MCET-V): MCET-V is a cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks
  Multiple Channel Exposure Therapy- Veterans: Individual therapy design completed twice a week over a 6-week period. The treatment will include psychoeducation about panic attacks and trauma and behavioral and cognitive exposure exercises.
Period: Overall Study
Arm/Group | Multiple Channel Exosure Therapy (MCET-V)
Started | 7
Completed | 2
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Multiple Channel Exposure Therapy (MCET): MCET-V is a cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks
  Multiple Channel Exposure Therapy- Veterans: Individual therapy design completed twice a week over a 6-week period. The treatment will include psychoeducation about panic attacks and trauma and behavioral and cognitive exposure exercises.
Arm/Group | Multiple Channel Exposure Therapy (MCET)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (6.9)
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Beck Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] — The Beck Anxiety Inventory (BAI) is a measure of general anxiety and consists of 21 items that are rated using a 4-point Likert scale ranging from 0 (not at all) to 3 (severely). The BAI ranges from a score of 0 to 63. Interpretation guidelines for the BAI are: 0-7 (minimal), 8-15 (mild), 16-25 (moderate), and 26-63 (severe).
  units on a scale | 40.6 (9.93)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory-II (BDI-II) is a measure of depression and consists of 21 items that are rated using a 4-point Likert scale ranging from 0 (little or no distress) to 3 (much distress). The BDI-II ranges from a score of 0 to 63. Interpretation guidelines for the BDI-II are: 0-13 (minimal), 14-19 (mild), 20-28 (moderate), and 29-63 (severe).
  units on a scale | 36.4 (8.11)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: The CAPS is a clinician-administered interview assessing 17 symptoms of PTSD (based on DSM-IV criteria). Frequency of symptoms are rated on a scale from 0 (never/none) to 4 (daily/almost every day). Intensity of symptoms are rated using a scale of 0 (none) to 4 (extreme). Total severity score is derived by summing the frequency and intensity scores. A recommended cut-off of 45 is used to determine the presence of full PTSD. Higher scores suggest greater symptom severity.
Time Frame: 1-week post-treatment (approximately week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MCET-V: MCET-V is a 12-session intervention targeting panic and PTSD symptoms.
Arm/Group | MCET-V
Number analyzed (Participants) | 2
units on a scale | 29.5 (23.3)

2. Secondary Outcome: Anxiety Disorders Interview Schedule- DSM-IV (ADIS-IV)
Description: The ADIS-IV is a semi-structured diagnostic interview for anxiety disorders (based on DSM-IV criteria). DSM-IV criteria for panic disorder include recurrent unexpected panic attacks and (1) persistant concern or worry about additional panic attacks or their consequences or (2) significant change in behavior related to panic attacks.
Time Frame: 3 Months
Measure: Number; unit: percentage of participants
Arm/Group | MCET-V
Number analyzed (Participants) | 2
percentage of participants
  Participants without panic disorder | 100
  Participants with panic disorder | 0

3. Primary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: 3-month follow-up (approximately week 26)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCET-V
Number analyzed (Participants) | 2
units on a scale | 17 (1.41)

ADVERSE EVENTS:
Groups:
- Arm 1: MCET-V is a cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks
  Multiple Channel Exposure Therapy- Veterans: Individual therapy design completed twice a week over a 6-week period. The treatment will include psychoeducation about panic attacks and trauma and behavioral and cognitive exposure exercises.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes